CLINICAL TRIAL: NCT00517400
Title: Evaluation of the H-Coil Transcranial Magnetic Stimulation (TMS) Device- Treatment for Post Traumatic Stress Disorder
Brief Title: Deep Transcranial Magnetic Stimulation (TMS)- Treatment for Post Traumatic Stress Disorder
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Moshe Isserles, MD, MSc, Hadassah Medical Organization
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 364/3.8.07(HMO)
Record Dates: First submitted 2007-08-16; First posted 2007-08-17 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2010-07

CONDITIONS: Post Traumatic Stress Disorder
Keywords: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (3):
- Exposure-Stimulation (Active Comparator)
  Interventions: Device: Deep repetitive Transcranial Magnetic Stimulation (rTMS) real or sham
- Sham exposure - Real stimulation (Active Comparator)
  Interventions: Device: Deep repetitive Transcranial Magnetic Stimulation (rTMS) real or sham
- Exposure - Sham Stimulation (Active Comparator)
  Interventions: Device: Deep repetitive Transcranial Magnetic Stimulation (rTMS) real or sham

INTERVENTIONS:
Device: Deep repetitive Transcranial Magnetic Stimulation (rTMS) real or sham
  Other Names: Brainsway H-Coil

SUMMARY:
Evaluation of the novel deep TMS H-Coil designs as a treatment measure in post traumatic stress disorder (PTSD).

Comparing real to sham treatment.

ELIGIBILITY:
Inclusion Criteria:

* PTSD diagnosis per DSM IV

Exclusion Criteria:

* Schizophrenia
* Bipolar I
* severe Axis II diagnosis
* risk factors to convulsions
* drug / alcohol abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-02; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
CAPS SCORE [TOTAL, INTRUSION] | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Isserles, MD, MSc, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Psychiatric department, Hadassah-Hebrew universityMedical Organization, Jerusalem, Israel

REFERENCES:
- [Result] Isserles M, Shalev AY, Roth Y, Peri T, Kutz I, Zlotnick E, Zangen A. Effectiveness of deep transcranial magnetic stimulation combined with a brief exposure procedure in post-traumatic stress disorder--a pilot study. Brain Stimul. 2013 May;6(3):377-83. doi: 10.1016/j.brs.2012.07.008. Epub 2012 Aug 18. PMID 22921765